CLINICAL TRIAL: NCT03503110
Title: Anatomo-functional Study of the Brain Cortical and Sub-cortical Connectivity Using Diffusion MRI, Electrocorticography and Direct Electrical Stimulation
Brief Title: Bridging Brain Structure and Function by Correlating Structural Connectivity, Cortico-Cortical Transmission and Direct Electro-Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-PP-15
Record Dates: First submitted 2018-03-20; First posted 2018-04-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tumor, Brain
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dMRI and electrocorticography (Experimental): Direct measurements of cortical electrical properties of patients operated on awake surgery for a brain tumor, using electrocorticography (ECoG), based on the dMRI tractography data previously acquired for each patient.
  Interventions: Other: electrocorticography with electrostimulation; Other: dRMI

INTERVENTIONS:
Other: electrocorticography with electrostimulation — The investigators aim to establish a relationship between dMRI SC measures, direct measures of electrical properties of the human brain cortex obtained with electrocorticography (ECoG), and response elicited by direct electrostimulation of the brain (DES)
Other: dRMI — The investigators aim to establish a relationship between dMRI SC measures, direct measures of electrical properties of the human brain cortex obtained with electrocorticography (ECoG), and response elicited by direct electrostimulation of the brain (DES)

SUMMARY:
Elucidating the structure-function relationship of the brain is one of the main open questions in neuroscience. The capabilities of diffusion MRI-based (dMRI) techniques to quantify the connectivity strength between brain areas, namely structural connectivity (SC), in combination with modalities such as electroencephalography (EEG) to quantify brain function have enabled advances in this field. However, so far the actual relationship between SC measures and measures of information transport between neuronal patches has not been determined. In this project, we aim to establish a relationship between dMRI SC measures, direct measures of electrical properties of the human brain cortex obtained with electrocorticography (ECoG), and response elicited by direct electrostimulation of the brain (DES). Ten patients operated on awake surgery for brain tumor removal will be included. First, a dMRI will be acquired prior to the surgery, in order to extract SC indices through probabilistic tractography. Then, intrasurgical cortico-cortical electrical measures will be obtained by ECoG electrodes positioned on the predefined cortical terminations of the designated bundles. These measures will be correlated to functional responses obtained during the cortical cartography, following the common DES procedure. The results of this multi-modal approach combining structure and function explorations of the brain should help to elucidate the relationship between non-invasive (dMRI) SC measures and cortico-cortical transmission properties (delays, transfer functions), and should boost the understanding of cognitive function as well as neurosurgical planning for the treatment of pathologies such as brain tumor resection and drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible at an awake surgery for a brain tumor resection
* Informed consent of the patient

Exclusion Criteria:

* Contraindication to MRI
* Withdrawal of the patient's consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Descriptive activity of brain with dMRI results | after the operation (1 month)
Descriptive functional responses elicited by the direct electrostimulation of the cortex. | after the operation (1 month)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sporns O. The human connectome: origins and challenges. Neuroimage. 2013 Oct 15;80:53-61. doi: 10.1016/j.neuroimage.2013.03.023. Epub 2013 Mar 23. PMID 23528922
- [Result] Duffau H. Stimulation mapping of white matter tracts to study brain functional connectivity. Nat Rev Neurol. 2015 May;11(5):255-65. doi: 10.1038/nrneurol.2015.51. Epub 2015 Apr 7. PMID 25848923
- [Result] Yamao Y, Matsumoto R, Kunieda T, Arakawa Y, Kobayashi K, Usami K, Shibata S, Kikuchi T, Sawamoto N, Mikuni N, Ikeda A, Fukuyama H, Miyamoto S. Intraoperative dorsal language network mapping by using single-pulse electrical stimulation. Hum Brain Mapp. 2014 Sep;35(9):4345-61. doi: 10.1002/hbm.22479. Epub 2014 Feb 24. PMID 24615889
- [Result] Bates E, Wilson SM, Saygin AP, Dick F, Sereno MI, Knight RT, Dronkers NF. Voxel-based lesion-symptom mapping. Nat Neurosci. 2003 May;6(5):448-50. doi: 10.1038/nn1050. No abstract available. PMID 12704393
- [Result] Szelenyi A, Bello L, Duffau H, Fava E, Feigl GC, Galanda M, Neuloh G, Signorelli F, Sala F; Workgroup for Intraoperative Management in Low-Grade Glioma Surgery within the European Low-Grade Glioma Network. Intraoperative electrical stimulation in awake craniotomy: methodological aspects of current practice. Neurosurg Focus. 2010 Feb;28(2):E7. doi: 10.3171/2009.12.FOCUS09237. PMID 20121442
- [Result] Leclercq D, Duffau H, Delmaire C, Capelle L, Gatignol P, Ducros M, Chiras J, Lehericy S. Comparison of diffusion tensor imaging tractography of language tracts and intraoperative subcortical stimulations. J Neurosurg. 2010 Mar;112(3):503-11. doi: 10.3171/2009.8.JNS09558. PMID 19747052